CLINICAL TRIAL: NCT06416514
Title: Construction and Empirical Study of Personalized Intervention Based on Health Portrait in Mild Behavioral Impairment
Brief Title: Personalized Interventions Via Health Portraits in Mild Behavioral Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yuanjiao Yan, Principal Investigator, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-177
Record Dates: First submitted 2024-01-16; First posted 2024-05-16 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Neurocognitive Disorders
Keywords: Mild behavioral impairment; Older adults; Personalized intervention; Health portrait; Neuropsychiatric symptoms
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with high social participation (Experimental): Patients with high social participation were more active in health management and monitoring due to their high social participation. NPS symptoms were monitored regularly for patients in the different groups, and personalized interventions were developed according to the development of NPS symptoms and patient preferences.
  Interventions: Other: Personalized intervention
- Patients with low social participation (Experimental): In the low social participation group, due to the low social participation of patients, their initiative to participate in health management and monitoring is also low. For the patients in the reorganized group, their self-confidence and enthusiasm to participate in activities are first enhanced through health education and health popularization, and NPS symptoms are regularly monitored, and personalized intervention measures are formulated according to the development of NPS symptoms and patient preferences.
  Interventions: Other: Personalized intervention

INTERVENTIONS:
Other: Personalized intervention — Personalized intervention means implementing multi-component non-pharmacological interventions based on different health profiles，such as art therapy, exercise therapy, cognitive therapy and other monotherapies. Usual care means care as routine.
  Other Names: Usual care

SUMMARY:
The incidence of MBI and the probability of progression to dementia are high. Early detection and intervention have important clinical significance to reduce the occurrence of dementia, delay the progression of dementia and promote healthy aging to active aging. The occurrence and development of NPS in MBI patients may be related to genetic and degenerative changes in the central nervous system. The evaluation of MBI patients is mainly based on neuropsychological tests, including NPS and cognitive function assessment. Landmark model is an effective tool for dynamic risk prediction of the progress of MBI. It can make dynamic prediction at different time points according to various existing measurement indicators of an individual and calculate the individual prediction probability, which is one of the best models for studying the outcome of disease at present. The Landmark model is applied to the elderly MBI population to study the influencing factors of normal aging, MBI and dementia and the probability of metastasis, which is a beneficial attempt to further advance the defense line of dementia. Personalized non-drug intervention is the preferred treatment for MBI, which mainly includes cognitive/emotional intervention, sensory stimulation, exercise therapy, etc. Currently, it is recommended to adopt diversified strategies to implement individualized precision treatment programs for patients. The hierarchical and classified health management of elderly MBI patients combined with health portrait technology is helpful to improve management efficiency and better meet the needs of personalized health management for the elderly.

DETAILED DESCRIPTION:
Combined with the current situation of relevant research at home and abroad, it can be seen that the research in this field still has the following limitations:First, as a population with a high incidence of dementia, there are many studies on the influencing factors of dementia in elderly MBI, but there is heterogeneity in research design and other aspects, and no studies have effectively integrated it. Therefore, determining the risk factors of MBI in the elderly is helpful for effective risk factor management in the early stage of dementia, which is of great significance for delaying the speed of MBI in the elderly and reducing the burden of family and society.Second, most current studies are cross-sectional studies or the development and testing of assessment tools, and few studies pay in-depth attention to the development and change of NPS, ignoring the possibility of reversal of MBI. Further understanding of the natural history of MBI and the influence of demography, environment, lifestyle and other related factors on the occurrence and development of MBI, and understanding the change law of the occurrence and development of MBI are of great importance to find the breakthrough point of early and effective intervention.Third, there is still a lack of management guidelines for MBI, and it is urgent to develop personalized non-drug interventions for MBI patients. "Human-centered" multiple personalized intervention is expected to improve NPS symptoms in MBI patients, reduce the occurrence of dementia, and delay the progression of dementia.Fourth, as an emerging technology, health portrait has made some progress in the management of chronic disease symptoms at home and abroad, but its application in the specific subdivision of chronic disease management in the elderly is still limited. The application of health portrait in the management of NPS symptoms in elderly MBI patients is a new exploration.Therefore, this study raises three research questions: First, what is the current situation of mild behavioral impairment in the elderly? What are the relevant factors? Second, what are the risk factors that affect the outcome of mild behavioral impairment in the elderly? What is the probability of metastasis between different states in elderly patients with mild behavioral impairment? Third, how to build a personalized program for elderly MBI patients in China based on user portraits? How scientific, feasible and safe is it?In view of the above research problems, this study first understood the status quo of mild behavioral impairment in the elderly and explored its related factors; Then, the prediction model of mild behavioral impairment in the elderly was constructed to explore the factors affecting its outcome and its transfer probability. Finally, a personalized intervention system for elderly patients with mild behavioral impairment based on health profiles was developed and tested. The significance of this study is that in the context of the rapid development of population aging, the increasing promotion of the strategy of healthy China and the national strategy of actively coping with population aging, the completion of this study is expected to clarify the development and change mechanism of MBI, provide new ideas and new methods for the management of MBI patients, and also provide new evidence for the prevention and treatment of dementia high-risk groups. This is a low-cost and efficient strategic choice to deal with the aging population and reduce the burden of dementia, and has a good scientific application prospect and practical significance.

ELIGIBILITY:
Inclusion Criteria:

* Meet the ISTAART diagnostic criteria for MBI;
* Age ≥60 years old;
* No obvious visual or hearing impairment;
* Have the ability of language communication, can complete the scale assessment.

Exclusion Criteria:

* Patients with severe physical diseases and unable to complete cognitive function screening;
* Patients with other neurological diseases and serious medical diseases that can cause brain dysfunction.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
General cognitive function | The intervention was conducted in September 2024, and the evaluation time was 0,3 months separately
  The Montreal Cognitive Assessment Scale, developed by Nasreddine in 2004 to assess participants' general cognitive function, covers eight areas of cognitive assessment, including visuospatial and executive function, naming, memory, attention, speech, abstraction, delayed recall, and orientation. The Changsha version of the Montreal Cognitive Assessment Scale was used in this study, and its Cronbach's α coefficient was 0.846, retest reliability was 0.974, and investigator reliability was 0.969. The score of the Montreal Cognitive Assessment Scale ranges from 0 to 30 points. The higher the score, the better the cognitive function of the study subjects. The illiterate group ≤13, the primary school group ≤19, and the junior high school and above group ≤24 can be judged as impaired cognitive function to correct the bias caused by education level

SECONDARY OUTCOMES:
Sleep condition | The intervention was conducted in September 2024, and the evaluation time was 0,3 months separately
  The Pittsburgh Sleep Quality Index, developed by Buysse equals in 1989, was used to evaluate the sleep status of the participants over the past month. The Pittsburgh Sleep Quality Index includes seven components: subjective sleep quality, sleep duration, sleep duration, sleep efficiency, sleep disorders, hypnotic drugs, and daytime function, with good internal consistency (Cronbach's α=0.83) and retest reliability (r=0.85). The cumulative score for each component of the Pittsburgh Sleep Quality Index Scale is the total score of the scale, ranging from 0 to 21, with a score of 0 to 3 for each component, with higher scores associated with poorer sleep quality
Social participation | The intervention was conducted in September 2024, and the evaluation time was 0,3 months separately
  The Social Support Rating Scale was used to assess participants' social participation. This study adopted the social support assessment compiled by domestic scholar Xiao Shuiyuan, which has good reliability and validity (Cronbach's α coefficient is 0.83). There are 10 items in the social support evaluation, including objective support, subjective support and social support utilization. The score ranges from 11 to 40 points. The higher the score of each dimension, the higher the degree of social support. It is generally believed that the total score of 20 is poor social support, 20-30 is general social support, and 30-40 is satisfactory social support
Dementia conversion rate | The intervention was conducted in September 2024, and the evaluation time was 0,3 months separately
  The Condensed Mental State Scale, developed by Folstein et al., is increasingly being used to screen patients for dementia, determine the severity of cognitive impairment, and determine dementia transition. The sensitivity and specificity of the concise mental State scale in the screening diagnosis of dementia are 80-90% and 70-80%. The scale covers cognitive areas such as orientation, memory, attention and computation, speech and visuospatial. The Condensed Mental State Scale ranges from 0 to 30 points. Dementia can be graded according to the Condensed Mental State Scale, with mild dementia scoring 21-26, moderate dementia 11-20, and severe dementia 0-10
Psychological symptoms | The intervention was conducted in September 2024, and the evaluation time was 0,3 months separately
  The Neuropsychiatric Scale (NPI) is also a suitable tool for assessing NPS in patients with MBI. The Neuropsychiatric Scale is a scale developed by Cummings et al. to assess NPS in dementia patients, including hallucinations, delusions, agitation/aggression, anxiety, depression, euphoria, loss, disinhibition, abnormal movement, appetite disorders, sleep and nocturnal behavior disorders. The Chinese version of neuropsychiatric scale has good reliability and validity with Cronbach's α coefficient of 0.851, bias coefficient of 0.83, and total retest reliability of 0.86. The neuropsychiatric scale is easy to use and provides a way for semi-structured interviews to distinguish symptoms of inhibition from symptoms of apathy. Neuropsychiatric scale patient scores ranged from 0-144, caregiver pain scores ranged from 0-60, the lower the score the better
Behaviour impairment | The intervention was conducted in September 2024, and the evaluation time was 0,3 months separately
  The Mild Behavioral Impairment checklist (MBI-Checklist) asseses subjects to assess the symptoms and severity of MBI and was developed by ISTAART after the publication of diagnostic criteria for MBI in 2016. The mild behavioral impairment Checklist, filled out by a family member or someone in the know, has five categories, including lack of motivation, emotional incoordination, impulse control disorders, social withdrawal, and perceptual or thinking abnormalities. The sensitivity and specificity of the mild behavioral impairment checklist were 86.96% and 86.00%. The mild behavioral Impairment Checklist scores range from 0 to 102, with the higher the total score, the higher the degree of mild behavioral impairment

CONTACTS AND LOCATIONS:
Overall Officials: Yuanjiao Yan, PhD, Study Director — Shengli clinical medical college of Fujian Medical university
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China